CLINICAL TRIAL: NCT03695848
Title: Prognostic Value of Diffusion Tensor Imaging and fMRI in Surgical Management of Cervical Myelopathy
Brief Title: Prognostic Value of DTI and fMRI of Cervical Myelopathy
Acronym: CSM
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 18-394
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2019-04

CONDITIONS: Cervical Myelopathy
Keywords: Cervical Myelopathy，Prognostication，Diffusion Tensor Imaging, fMRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MRI scan — Before decompresssion surgery, DTI and fMRI will be recorded by a FDA approved 3T MRI scanner (Philips Achieva)

SUMMARY:
Cervical myelopathy (CM) is one of the most common degenerative spinal cord disorders affecting older people. The progression of CM is insidious and the neurological decline can vary between patients. Surgical decompression is considered the most effective way to treat CM, however, it is not free from risk and the surgical outcome is not always satisfactory. The expected outcome of surgical intervention for CM remains a difficulty. There is a pressing need for a reliable and quantitative approach to predict surgical outcomes of CM and the precise prognosis. Previous studies have suggested a number of prognostic factors, such as age, duration of symptoms, pre-operative neurological status and abnormal MRI, but their prognostic value remains controversial. Recently, diffusion tensor imaging (DTI) and fMRI have been proposed as a promising tool for predicting the surgical prognosis of CM. In previous study, the protocol was successfully established for DTI microstructural characterization and resting state fMRI of the cervical spinal cord. This study is to evaluate the value of DTI and fMRI in predicting the outcome of surgical treatment. The ultimate goal is to establish a clinical protocol for quantitative DTI and fMRI analysis that could give accurate prognosis for surgical intervention to CM.

DETAILED DESCRIPTION:
Cervical myelopathy (CM) is the most common cause of spinal cord dysfunction in the elderly. Symptoms often develop insidiously and are characterized by neck stiffness, arm pain, numbness in the hands, and weakness of the hands and legs. The causes of this myelopathy are many, such as spinal canal narrowing, osteophytes, herniated discs and hypertrophy of the ligamentum flavum. Although the clinical signs and symptoms of CM are well documented in the literature, a precise localization of the maximum level of compression is sometimes difficult in the elderly patients where multiple levels of the cervical spine are degenerated. Also the lack of understanding of the pathophysiology and pathomechanism of CM has significantly hampered the development of a rational approach to the surgical treatment of such condition.

The diagnosis is made based on clinical signs and symptoms with the help of conventional MRI imaging which demonstrates the levels of anatomical stenosis. Surgical decompression of the cervical spine is the most common form of treatment. Magnetic resonance imaging (MRI) has been used widely in the evaluation of patients with CM. The commonly applied MR techniques include spin echo sequence, both conventional spin echo and fast/turbo spin echo for T1 and T2 information; gradient echo sequences, which generate T2 images; STIR (short tau inversion recovery) images; fat suppressed T1 images; gadolinium enhanced images applied to either routine T1WIs or fat suppressed T1WIs; MR spinal angiography; and cerebrospinal fluid flow (CSF) studies (either magnitude or phase contrast). However, conventional MRI mainly concerns anatomical information about CM, with less pathophysiological information. BOLD-fMRI is able to present the activated neuronal volume decreased in CM patients along with an increase in neuronal activities. diffusion tensor imaging (DTI) permits the detection of tissue-water molecular diffusion at microscopic dimensions. Previous studies have demonstrated the feasibility of DTI in evaluating microstructural changes in the myelopathic cervical cord. The prognostic values of spinal cord DTI in CM have been addressed in several previous studies. In recent years, combination of DTI and fMRI has been proposed to be an accurate prognostic tool for surgical management of CM.

Cervical myelopathy (CM) is caused by degenerative stenosis of the cervical spine with progressive compression on the spinal cord resulting in loss of sensory and motor functions in the upper and lower limbs. Surgical decompression of the cervical spine is the most common form of treatment.

The objective of this project is to evaluate the value of DTI and fMRI in predicting the outcome of surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are a clinical diagnosis of CM including the signs of corticospinal lesions together with the appropriate radiographic findings.

Exclusion Criteria:

* Patients with acute spinal cord injuries, prior spinal intervention, with shrapnel or other metal or electronic implants in their bodies (such as pacemakers, aneurysm clips, surgical devices, metallic tattoos on the head, etc.), with claustrophobia and pregnant women will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical myelopathy requiring surgical decompression will be recruited.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative neurological improvement rate | Baseline on enrollment and 12 months follow-up
  comparison of clinical spinal cord functional changes between pre- and post-operative status.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - G Li, Hong Kong
  - The university of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No